CLINICAL TRIAL: NCT02089035
Title: Replacement of Saturated Fat in Dairy on Total Cholesterol, Vascular Function, Ambulatory Blood Pressure and Cardiovascular Risk Biomarkers
Brief Title: Replacement of Saturated Fat in Dairy on Total Cholesterol
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 13/43; University of Reading (Other: University of Reading)
Record Dates: First submitted 2014-01-05; First posted 2014-03-17 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2016-05

CONDITIONS: Hypercholesterolemia
Keywords: Milk fatty acids; Total cholesterol; Vascular function; Blood pressure
MeSH Terms: conditions — Hypercholesterolemia | interventions — Cheese; Butter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MUFA-rich dairy products (Experimental): Subjects are asked to exchange habitual dairy products for modified MUFA-rich experimental dairy products for a 12 week period.
  Participants will provided with standardised quantities of pasteurised UHT milk, cheese and butter that they will be asked to consume on a daily basis.
  Interventions: Dietary Supplement: MUFA-rich dairy products (UHT milk, cheese and butter)
- Conventional dairy products (Experimental): Subjects are asked to consume habitual non-modified dairy products for a period of 12 weeks.
  Participants will provided with standardised quantities of pasteurised UHT milk, cheese and butter that they will be asked to consume on a daily basis.
  Interventions: Dietary Supplement: Conventional dairy products (UHT milk, cheese, butter)

INTERVENTIONS:
Dietary Supplement: MUFA-rich dairy products (UHT milk, cheese and butter)
  Arms: MUFA-rich dairy products
Dietary Supplement: Conventional dairy products (UHT milk, cheese, butter)
  Arms: Conventional dairy products

SUMMARY:
The consumption of milk and dairy products is recognised as an essential part of a healthy diet as it represents an important source of key micro- and macronutrients. Nevertheless, there is still a widespread conviction that the overall high energy density and concentration of long-chain saturated fatty acids (SFA) present in dairy have detrimental health effects, contributing to the progression of cardiovascular disease, obesity and diabetes.

Supplementation of the bovine diet with a source of MUFA, such as rapesee oil, has become an achievable strategy in order to reduce the amount of SFA present in dairy products.

The aim of this project is to observe the effects of three types of dairy products (UHT milk, cheese and butter) produced from milk derived from cows fed withhigh-oleic sunflower oil, on CVD risk biomarkers and plasma total cholesterol levels in adults with an increased risk of developing CVD. The aim is to determine whether an isoenergetic exchange of dairy products will affect vascular function and CVD biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mildly hypercholesterolemic: TC <5.2 and <8mmol/L
* Age: 25-70
* BMI: 19-32 kg/m2
* Haemoglobin: >125g/L for women and 135g/L for men
* Normal liver and kidney function

Exclusion Criteria:

* Milk, cheese, butter, lactose allergy
* Drug treatment for hyperlipidaemia, hypertension, inflammation and hypercoagulation
* Suffered myocardial infarction/stroke in the past 12months
* Diabetic (diagnosed or fasting glucose > 7 mmol/l) or suffer from other endocrine disorders
* Surgery in the previous 6 months
* Excessive alcohol consumption (>28 unit/wk man; >21 unit/wk women)
* Taking vitamin, mineral or fatty acid supplements (e.g. fish oil, calcium)
* Pregnant, lactating, planning a pregnancy or not using effective contraceptive precautions
* Smokers
* Vegans
* Anaemic
* Planning or on a weight reduction scheme
* Parallel participation in another intervention study
* Participating in intensive aerobic activity for > 20 minutes 3 times per week
* Use of anti-inflammatory medication

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Chronic study: Changes in fasting plasma circulating levels of total cholesterol | Chronic study: Baseline and week 12 for both intervention arms
Acute study: Changes in postprandial flow-mediated dilatation | Acute study: 0, 180, 300 and 420 min at baseline and week 12 for both intervention arms

SECONDARY OUTCOMES:
Changes in vascular stiffness by Carotid Intima Media Thickness (CIMT) | Chronic study: Baseline measurements (0min) for both intervention arms
Change in 24-hour ambulatory blood pressure | Chronic study: baseline (-1week) and week 11, 19 and 31 for 24 hours. Measurements will be recorded every 30min (7am to 10pm) and every hour (10pm-7am)
Changes in plasma circulating markers of vascular health | Chronic study: Baseline and week 12 for both intervention arms. Acute study: area under the curve from 0-8 h after consumption of breakfast (0 min) and lunch (330 min) for both intervention arms
Changes in plasma circulating markers of inflammatory status | Chronic study: Baseline and week 12 for both intervention arms. Acute study: area under the curve from 0-8 h after consumption of breakfast (0 min) and lunch (330 min) for both intervention arms
Changes in plasma circulating markers related to lipid metabolism | Chronic study: Baseline and week 12 for both intervention arms. Acute study: area under the curve from 0-8 h after consumption of breakfast (0 min) and lunch (330 min) for both intervention arms
Changes in plasma circulating markers related to insulin resistance | Chronic study: Baseline and week 12 for both intervention arms. Acute study: area under the curve from 0-8 h after consumption of breakfast (0 min) and lunch (330 min) for both intervention arms
Changes in vascular stiffness by Pulse Wave Velocity (PWV) | Chronic study: Baseline (0 min) and week 12 for both intervention arms
Changes in vascular stiffness by Pulse Wave Analysis (PWA) | Chronic study: Baseline (0 min) and week 12 for both intervention arms
Changes in vascular stiffness by Digital Volume Pulse (DVP) | Chronic study: Baseline (0 min) and week 12 for both intervention arms
Changes in monocytic cytokine production from whole blood culture | Chronic and acute study: Baseline and week 12 for both intervention arms. Acute: area under the curve from 0-8 h following consumption of breakfast (0 min) and lunch (330 min) for both intervention arms
Changes in vascular reactivity by Flow Mediated Dilatation (FMD) | Chronic study: Baseline and assessment at 12 weeks for each intervention arm.
Changes in anthropometric measurements | Chronic study: Baseline and assessment at 12 weeks for each intervention arm.
Change in plasma phospholipid fatty acid composition | Chronic and acute study: Baseline and week 12 for both intervention arms. Acute study: 0, 180, 300 and 420 min at baseline and week 12 for both intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berks, United Kingdom

REFERENCES:
- [Background] Livingstone KM, Lovegrove JA, Givens DI. The impact of substituting SFA in dairy products with MUFA or PUFA on CVD risk: evidence from human intervention studies. Nutr Res Rev. 2012 Dec;25(2):193-206. doi: 10.1017/S095442241200011X. Epub 2012 Aug 6. PMID 22863409
- [Background] Elwood PC, Pickering JE, Givens DI, Gallacher JE. The consumption of milk and dairy foods and the incidence of vascular disease and diabetes: an overview of the evidence. Lipids. 2010 Oct;45(10):925-39. doi: 10.1007/s11745-010-3412-5. Epub 2010 Apr 16. PMID 20397059
- [Derived] Markey O, Vasilopoulou D, Kliem KE, Fagan CC, Grandison AS, Sutton R, Humphries DJ, Todd S, Jackson KG, Givens DI, Lovegrove JA. Postprandial Fatty Acid Profile, but Not Cardiometabolic Risk Markers, Is Modulated by Dairy Fat Manipulation in Adults with Moderate Cardiovascular Disease Risk: The Randomized Controlled REplacement of SaturatEd fat in dairy on Total cholesterol (RESET) Study. J Nutr. 2021 Jul 1;151(7):1755-1768. doi: 10.1093/jn/nxab050. PMID 33758921
- [Derived] Vasilopoulou D, Markey O, Kliem KE, Fagan CC, Grandison AS, Humphries DJ, Todd S, Jackson KG, Givens DI, Lovegrove JA. Reformulation initiative for partial replacement of saturated with unsaturated fats in dairy foods attenuates the increase in LDL cholesterol and improves flow-mediated dilatation compared with conventional dairy: the randomized, controlled REplacement of SaturatEd fat in dairy on Total cholesterol (RESET) study. Am J Clin Nutr. 2020 Apr 1;111(4):739-748. doi: 10.1093/ajcn/nqz344. PMID 32020168
- [Derived] Markey O, Vasilopoulou D, Kliem KE, Koulman A, Fagan CC, Summerhill K, Wang LY, Grandison AS, Humphries DJ, Todd S, Jackson KG, Givens DI, Lovegrove JA. Plasma phospholipid fatty acid profile confirms compliance to a novel saturated fat-reduced, monounsaturated fat-enriched dairy product intervention in adults at moderate cardiovascular risk: a randomized controlled trial. Nutr J. 2017 May 23;16(1):33. doi: 10.1186/s12937-017-0249-2. PMID 28535777